CLINICAL TRIAL: NCT00657397
Title: Initialization of Methadone in Primary Care; a Randomized Intervention Research for Preventing HCV Transmission Practices. ANRS Methaville
Brief Title: Initialization of Methadone in Primary Care, Randomized Intervention Research for Preventing HCV Transmission Practices
Acronym: Methaville
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: French National Agency for Research on AIDS and Viral Hepatitis (Other Government)
Responsible Party: Sponsor
Organization: ANRS, Emerging Infectious Diseases (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS Methaville
Record Dates: First submitted 2008-04-08; First posted 2008-04-14 (Estimated); Last update posted 2012-07-24 (Estimated); Status verified 2012-07

CONDITIONS: Hepatitis C; Substance Dependence; Methadone
Keywords: Methadone; Substance Dependence
MeSH Terms: conditions — Hepatitis C; Substance-Related Disorders | interventions — Methadone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Methadone inducted by a primary care physician
  Interventions: Drug: Methadone
- B (Active Comparator): Methadone inducted (in CSAPA)
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Methadone — Methadone sirup once daily

SUMMARY:
The rapid scale up of opioid substitution treatment (OST) for drug users mainly achieved through the possibility of prescribing buprenorphine in primary care has been successful in reducing HIV prevalence among drug users but still inadequate for reducing the spread of HCV. To date, methadone in France can only be initialised in drug centres but GPs can prescribe methadone after stabilisation of dosages.

This study was born as an answer to a request from the French Minister of Health that supports the initialisation of methadone in primary care in order to improve coverage by OST (now 70%) in drug users.

DETAILED DESCRIPTION:
We aimed to test the non inferiority of the proportion of non users of street-opioids after one year of treatment in patients inducted in primary care (PC) vs.those inducted in a specialised center for substance dependence (CSAPA).

In this multisite, open-label, randomised controlled non-inferiority trial, opioid dependent individuals were randomized to start methadone either in PC or in a CSAPA. After stabilization of methadone dosage (~2 weeks), patients could change arm. Follow-up assessments through medical questionnaires and phone interviews was scheduled at month 0 (M0, enrolment) M3, M6, M12. The opiate treatment index (OTI) was used for computing the proportion of patients reporting no use of street opioids in the last month at M12 (primary outcome) in those inducted in PC or in a CSAPA and the non inferiority margins.

Primary analysis was by intention to treat (ITT)

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 years patients needing methadone for their opioid dependence who are either naives of methadone treatment (prescribed) since at least 1 month
* need to switch from buprenorphine to methadone treatment
* negative test for pregnancy

Exclusion Criteria:

* co-dependent on alcohol and benzodiazepines,
* inmates,
* pregnant women,
* individual in irregular situation or who cannot be joined by phone.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 197 (Actual)
Dates: Start 2009-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
prevalence of non-users of street opioid after one year of treatment will be compared between arms. | one year

SECONDARY OUTCOMES:
Prevalence of non users of street opioids after three months of treatment | three months
Retention in treatment | one year
Decrease in HCV risk behaviors, addictive behaviors, improvement in quality of life, psychiatric comorbidities, social insertion, reduction in criminal acts | one year
cost-effectiveness | one year
surveillance of severe adverse events and overdose cases in each arm | Day -7 to Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Alain Morel, MD, Principal Investigator — CSST Le trait d'union, 154 rue du vieux pont de Sèvres, 92100 Boulogne, France; Patrizia Carrieri, PHD, Study Director — ORS PACA - INSERM-IRD UMR912, 23, rue Stanislas Torrents, 13006 Marseille
Locations (1):
- CSST Le trait d'union, Boulogne, France

REFERENCES:
- [Derived] Perry D, Kirkwood JE, Doroshuk ML, Kelmer M, Korownyk CS, Ton J, Garrison SR. Opioid agonist therapy for opioid use disorder in primary versus specialty care. Cochrane Database Syst Rev. 2025 Sep 8;9(9):CD013672. doi: 10.1002/14651858.CD013672.pub2. PMID 40919724
- [Derived] Carrieri P, Vilotitch A, Nordmann S, Lions C, Michel L, Mora M, Morel A, Maradan G, Spire B, Roux P; Methaville Study Group. Decrease in self-reported offences and incarceration rates during methadone treatment: A comparison between patients switching from buprenorphine to methadone and maintenance treatment incident users (ANRS-Methaville trial). Int J Drug Policy. 2017 Jan;39:86-91. doi: 10.1016/j.drugpo.2016.08.005. Epub 2016 Oct 19. PMID 27770695
- [Derived] Roux P, Lions C, Vilotitch A, Michel L, Mora M, Maradan G, Marcellin F, Spire B, Morel A, Carrieri PM; ANRS Methaville study group. Correlates of cocaine use during methadone treatment: implications for screening and clinical management (ANRS Methaville study). Harm Reduct J. 2016 Apr 5;13:12. doi: 10.1186/s12954-016-0100-7. PMID 27048152
- [Derived] Carrieri PM, Michel L, Lions C, Cohen J, Vray M, Mora M, Marcellin F, Spire B, Morel A, Roux P; Methaville Study Group. Methadone induction in primary care for opioid dependence: a pragmatic randomized trial (ANRS Methaville). PLoS One. 2014 Nov 13;9(11):e112328. doi: 10.1371/journal.pone.0112328. eCollection 2014. PMID 25393311
- [Derived] Roux P, Lions C, Michel L, Mora M, Daulouede JP, Marcellin F, Spire B, Morel A, Carrieri PM; ANRS Methaville study group. Factors associated with HCV risk practices in methadone-maintained patients: the importance of considering the couple in prevention interventions. Subst Abuse Treat Prev Policy. 2014 Sep 10;9:37. doi: 10.1186/1747-597X-9-37. PMID 25209306
- [Derived] Lions C, Carrieri MP, Michel L, Mora M, Marcellin F, Morel A, Spire B, Roux P; Methaville Study Group. Predictors of non-prescribed opioid use after one year of methadone treatment: an attributable-risk approach (ANRS-Methaville trial). Drug Alcohol Depend. 2014 Feb 1;135:1-8. doi: 10.1016/j.drugalcdep.2013.10.018. Epub 2013 Oct 31. PMID 24268548
- [Derived] Roux P, Michel L, Cohen J, Mora M, Morel A, Aubertin JF, Desenclos JC, Spire B, Carrieri PM; ANRS Methaville Study Group. Methadone induction in primary care (ANRS-Methaville): a phase III randomized intervention trial. BMC Public Health. 2012 Jun 28;12:488. doi: 10.1186/1471-2458-12-488. PMID 22741944